CLINICAL TRIAL: NCT01150942
Title: A Multi-center, Active-control, Randomized, Double-blind Phase 3 Clinical Trial to Assess the Immunogenicity and Safety of the Vero Cell-derived Inactivated Japanese Encephalitis Vaccine 'KD-287(JEIMMUGEN INJ.) in Korean Healthy Children Aged 12~23 Months
Brief Title: Clinical Trial to Assess the Immunogenicity and Safety of the Vero Cell-derived JE Vaccine in Korea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Seoul National University Hospital (Other); Gachon University Gil Medical Center (Other); Inha University Hospital (Other); Inje University (Other); Korea Cancer Center Hospital (Other); Samsung Medical Center (Other); The Catholic University of Korea (Other); Ewha Womans University (Other); Wonju Severance Christian Hospital (Other); Kyunghee University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KD287-BR-CT-301
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2011-02

CONDITIONS: Japanese Encephalitis
Keywords: JEV; vero cell
MeSH Terms: conditions — Encephalitis, Japanese | interventions — SA-14-14-2 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vero cell-derived JE vaccine (Experimental): vero cell-derived vaccine group
  Interventions: Biological: JE vaccine
- Mouse brain-derived JE vaccine (Active Comparator): Mouse brain-derived JE vaccine group
  Interventions: Biological: JE vaccine

INTERVENTIONS:
Biological: JE vaccine — 3 times, IM

SUMMARY:
To assess the immunogenicity and safety of the vero cell-derived inactivated JE vaccine in Korean healthy children aged 12~23 months

DETAILED DESCRIPTION:
To compare the Vero cell-derived inactivated Japanese encephalitis(JE) vaccine 'KD-287(JEIMMUGEN INJ.)' with the mouse brain-derived inactivated JE vaccine in terms of the immunogenicity and safety, in Korean healthy children aged 12~23 months

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 12-23 months
* Written informed consent

Exclusion Criteria:

* History of documented HIV
* Known or suspected impairment of immunologic function
* History of serious chronic disease
* Received any JE vaccine prior to enrollment

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 205 (Actual)
Dates: Start 2010-08; Primary Completion 2012-09 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
immunogenicity | pre-dose, after 3rd vaccination
  the seroconversion rates for JE antibodies 4 weeks after 3rd vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Hoan Jong Lee, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Yun KW, Lee HJ, Kang JH, Eun BW, Kim YJ, Kim KH, Kim NH, Hong YJ, Kim DH, Kim HM, Cha SH. Safety and immunogenicity of a freeze-dried, Vero cell culture-derived, inactivated Japanese encephalitis vaccine (KD-287, ENCEVAC(R)) versus a mouse brain-derived inactivated Japanese encephalitis vaccine in children: a phase III, multicenter, double-blinded, randomized trial. BMC Infect Dis. 2015 Jan 8;15:7. doi: 10.1186/s12879-014-0744-4. PMID 25567119